CLINICAL TRIAL: NCT06526351
Title: Immediate Vs. Conventional Loading for Early Implant Placement in the Esthetic Zone of Maxilla: Randomized Controlled Clinical Trial
Brief Title: Immediate vs Conventional Loading for Early Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Principal Investigator, Aleksa Markovic, Professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36/2
Record Dates: First submitted 2024-07-16; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Dental Implant
Keywords: early implant placement; immediate provisionalization

STUDY DESIGN:
Intervention Model Description: The study is designed as a single center, double-blinded, randomized, patient-oriented, controlled clinical trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Early implant placement + immediate provisionalization) (Experimental): Patients in test group receive an implant 6 to 8 weeks following tooth extraction with immediate provisional restoration
  Interventions: Device: Early implant placement with immediate provisional restoration
- Control group (Early implant placement + delayed loading) (Active Comparator): Patients in control group receive an implant 6 to 8 weeks following tooth extraction with submerged healing and conventional loading
  Interventions: Device: Early implant placement with delayed loading

INTERVENTIONS:
Device: Early implant placement with immediate provisional restoration — Implants placed following early implant placement protocol with soft tissue healing (6-8 weeks after tooth extraction). GBR procedure performed together with implant placement. Immediate provisional restoration will be delivered.
  Arms: Test group (Early implant placement + immediate provisionalization)
Device: Early implant placement with delayed loading — Implants placed following early implant placement protocol with soft tissue healing (6-8 weeks after tooth extraction). GBR procedure performed together with implant placement. Delayed loading protocol followed.
  Arms: Control group (Early implant placement + delayed loading)

SUMMARY:
The goal of this study is to assess clinical, radiological and patient centred outcomes of immediate and conventional implant loading protocols, and to compare clinical outcomes of these two different loading protocols (immediate and conventional) in combination with early implant placement of single implants in the esthetic zone of maxilla.

DETAILED DESCRIPTION:
Patients with a single failing tooth in the esthetic zone of maxilla (second premolar to second premolar), and in need for implant replacement will be recruited.

During the first appointment, medical history and clinical and radiological evaluations (OPG) will be recorded to verify the eligibility of each subject. If the sufficient bone is present apical to the failing tooth, intraoral scan of the upper jaw will be obtained prior to tooth extraction. Six to eight weeks following tooth extraction CBCT scan will be obtained together with digital impression. The implant positions will be planned according to the bone anatomy and future prosthetic reconstruction. Two groups of treatment protocols will be randomized as following:

Group 1: Early implant placement + immediate provisionalisation; Group 2: Early implant placement + conventional loading.

Implant surgery will be performed by two experienced surgeons. Full thickness triangular flap will be elevated, and fully guided implant placement will be completed. Under-preparation of implant bed in the soft bone will be utilized to obtain adequate primary stability. During the surgery, primary implant stability will be monitored by the means of insertion torque (IT) and resonance frequency analysis (RFA) Contour augmentation will be done for all patients from both groups by means of locally collected autogenous bone chips and deproteinized bovine bone particles, covered by a collagen membrane. Depending on the group, healing cap or healing abutment will be selected, and primary wound closure will be achieved.

Prosthetic rehabilitation:

All impressions will be taken digitally using intraoral scanner and appropriate implant scanbody.

Titanium temporary abutments will be used for provisional restorations, and titanium base abutments for the definitive restoration. Provisional restorations will be made of polymethyl methacrylate (PMMA) (Telio®CAD, Ivoclar Vivadent, Schaan, Lichtenstein) in a digital way. Digital scanning for final restorations and virtual design will be repeated in the same manner. Full ceramic screw-retained crown will be fabricated in a digital way and delivered to the patients.

Group 1:

Immediate screw-retained provisional restoration made of poly methyl methacrylate (PMMA) will be delivered within the first 7 days after surgery. Three months later, final screw-retained full ceramic crown will be fabricated and delivered.

Group 2:

Three months after the surgery, implant will be exposed and provisional screw-retained PMMA restoration delivered. Three months later final screw-retained ceramic crown will be fabricated.

Implant stability will be monitored through RFA. ISQ will be measured in both groups:

* At the day of the implant placement
* At the day of the provisional restoration placement
* At the day of the definitive restoration placement

CBCT scan with a small field of view will be taken prior to implant placement, immediately after implant placement, and 1 year after implant placement. Post-op CBCT scans will be used for measurement of the facial bone wall thickness. Marginal bone level will be monitored using periapical radiographs taken with paralleling technique, using custom silicone holder fabricated for each patient. X-rays will be taken on the day of the provisional restoration placement, final restoration placement, and one year after final restoration.

Esthetic outcome for the peri-implant mucosa will be assessed from the photographs taken at the definitive restoration delivery and 1 year follow-up visit, using pink esthetic score (PES). Patient satisfaction regarding function and aesthetics (mucosa, crown and overall) would be assessed using visual analogue scale (VAS). Quality of life would be examined by OHIP-14 questionnaire. These Patient Reported Outcome Measures (VAS and OHIP-14) would be recorded at 3 time points: before implant placement (baseline), 1 month after definitive crown delivery and after 1 year of function.

ELIGIBILITY:
Inclusion Criteria:

* Single failing tooth in the esthetic zone of maxilla (second premolar to second premolar)
* Patients older than 18 years
* Healthy patients ASA I and II
* Non-smokers/Light smokers (<10 cigarettes per day)
* Adequate bone volume apical and palatal to the failing tooth to allow for sufficient primary - implant stability of regular diameter implant

Exclusion Criteria:

* Implants adjacent to the failing teeth
* Active periodontal infection
* Severe bruxism
* Systemic or local conditions that contraindicates dental implant surgery - Heavy smokers (>10 cigarettes per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Marginal bone level changes | 1 year
  Marginal bone level will be monitored using periapical radiographs taken with paralleling technique, using custom silicone holder fabricated for each patient. X-rays will be taken on the day of the provisional restoration placement, final restoration placement, and one year after final restoration.
Pink esthetic score | 1 year
  Esthetic outcome for the peri-implant mucosa will be assessed from the photographs taken at the definitive restoration delivery and 1 year follow-up visit. Seven variables (mesial papilla, distal papilla, soft-tissue level, soft- tissue contour, alveolar process deficiency, soft-tissue color and texture) are assessed with a score 0, 1 or 2. Highest possible score is 14.

SECONDARY OUTCOMES:
Implant survival | 1 year
  Implant survival is assessed at provisional restoration delivery, final restoration delivery and at 1 year follow up
Facial bone wall width | 1 year
  Facial bone wall width is measured in mm at CBCT scans obtained immediately after implant placement and 1 year after final restoration delivery
Alveolar ridge volume | 1 year
  Alveolar ridge volume changes will be measured in mm in the image analysis software , by superimposing digital models (STL files) obtained prior to tooth extraction, prior to implant placement, at final restoration delivery, and 1year after final restoration delivery.
Patient satisfaction | 1 year
  Patient satisfaction regarding function and aesthetics (mucosa, crown and overall) would be assessed using visual analogue scale (VAS). It is recorded in 4 time points: before tooth extraction, before implant placement, 1 month after definitive crown delivery and after 1 year of function.
Impact of oral health on patient's quality of life | 1 year
  Oral Health Impact Profile (OHIP-14) questionnare will be used. Patients will fill a questionnare of 14 questions with responses made on a 5-point scale, coded 0 (never), 1 (hardly ever), 2 (occasionally), 3 (fairly often), and 4 (very often). Scores can range from 0 to 56, with higher OHIP-14 scores indicating worse and lower scores indicating better oral health related quality of life. It is recorded in 4 time points: before tooth extraction, before implant placement, 1 month after definitive crown delivery and after 1 year of function.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksa Markovic, Professor, Principal Investigator — Chair of Implant Center, School of Dental Medicine
Locations (1):
- Implant Center, School of Dental Medicine, Univeristy of Blegrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No